CLINICAL TRIAL: NCT05424666
Title: The Role of Lipofilling After Oncoplastic Breast Surgeries : Evaluation of Outcomes and Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mina rashad helmy besada, Assiut lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Oncoplastic breast surgeries
Record Dates: First submitted 2021-12-27; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient going Oncoplastic Breast surgeries (Experimental): Lipofilling After Oncoplastic Breast surgeries : Evaluation of Outcomes and Patient Satisfaction
  Interventions: Procedure: Harvesting method and Fat graft preparation method

INTERVENTIONS:
Procedure: Harvesting method and Fat graft preparation method — The procedure begins by identifying the areas where the fat will be collected Then the sample is collected by micro-incision using a fine suction cannula or during conventional liposuction. The fat cells are taken from an area of the body where there is a reserve (generally, in the abdomen, hips, knees, inner thighs, buttock) The collected fat cells are then subjected to a sterile centrifugation for a few minutes so as to separate the cells that will be injected (intact fat cells) from the elements that must not be injected (fat cells destroyed by the sample, non-fat cells such as than blood cells).
  Injection of fat cells into the breasts The reinjection of fat (lipofilling) is performed using micro-cannulas allowing incisions of the order of 1-2 mm in different angles and in multiple directions so as to increase the contact area between the grafted cells and the recipient tissues allowing a "good grip" of the injection.

SUMMARY:
The Role of Lipofilling After Oncoplastic Breast surgeries : Evaluation of Outcomes and Patient Satisfaction

DETAILED DESCRIPTION:
Lipofilling is the process of relocating autologous fat to change the shape, volume, consistency and profile of tissues. For over a century, surgeons have used autologous fat to enlarge and reshape the breasts.

Autologous fat grafting has gained popularity in recent years, although concerns exist regarding the safety and efficacy of this practice in breast surgery . Autologous fat grafting represents an important tool for the management of secondary contour deformities of reconstructed breasts; fat grafting is a simple, safe, and effective treatment option, with low morbidity. it is a straightforward and quick reconstructive technique that does not generally interfere with adjuvant therapies .patient surveys have demonstrated that irradiation has a significant and negative effect on patient satisfaction . Fat grafting seems to reduce radiation induced complications .improve cosmetic results, and reduce postoperative discomfort and pain. The aim of this study is to measure patient satisfaction with their breasts, as well as quality of life.

With the advent of liposuction in the 1980s, large amounts of unwanted fat could be removed from different body areas using small access incisions and a suction cannula. In this setting, fat grafting was re-introduced in the early 80s, pioneered by the American Mel Bircoll, who first described a series of fat transplantation for breast augmentation and reconstruction

ELIGIBILITY:
Inclusion Criteria:

Female gender.

Age of 18 years and older.

History or in candidate for a mastectomy in the near future.

Patients undergoing prophylactic mastectomy.

Patients' choice to undergo a breast reconstruction.

Wanting to participate in this study.

Patient is able to wear the BRAVA (BRA like VAcuum-based external tissue expander) device.

Exclusion Criteria:

Active smoker or a history of smoking 4 weeks prior to surgery.

Current substance abuse.

History of lidocaine allergy.

Four weeks or less after chemotherapy.

History of radiation therapy in the breast region.

Oncological treatment includes radiotherapy after mastectomy.

Kidney disease.

Steroid dependent (daily or weekly).

Immune-suppressed or immune-compromised disease.

Uncontrolled diabetes.

body mass index of >30.

Large breast size (ie, larger than cup C), unless the patient prefers reduction of the contralateral side towards cup C.

Extracapsular silicone leaking from the encapsulated implant from a previous breast reconstruction.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-19 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Cosmetic apperance | 1 week
  Volumetric evaluation of breast after surgery and symmetry to the other breast

SECONDARY OUTCOMES:
Complications during the treatment and follow up | 1 month
  Complications during the treatment Follow-up period will be registered and compared between the intervention and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Age / sex / clincal diagnosis
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: Assiut university